CLINICAL TRIAL: NCT05192460
Title: A Dose-Escalation and Dose-Expansion Study Evaluating the Safety and Efficacy of Personalized Neoantigen Vaccine in Advanced Gastric Cancer, Esophageal Cancer and Liver Cancer
Brief Title: Safety and Efficacy of Personalized Neoantigen Vaccine in Advanced Gastric Cancer, Esophageal Cancer and Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: jianming xu (Other)
Collaborators: NeoCura (Industry)
Responsible Party: Sponsor-Investigator, jianming xu, Principal Investigator, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKY- 1005
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Gastric Cancer; Esophageal Cancer; Liver Cancer
Keywords: Vaccine; Neoantigen
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: single-center, open-label, single-arm exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoantigen tumor vaccine with or without PD-1/L1 (Experimental): In dose escalation phase, subject will only receive neoantigen tumor vaccine. In dose expansion phase, subject will receive neoantigen tumor vaccine combination with PD-1/L1.
  Interventions: Biological: neoantigen tumor vaccine with or without PD-1/L1

INTERVENTIONS:
Biological: neoantigen tumor vaccine with or without PD-1/L1 — In dose escalation phase, subjects will receive neoantigen tumor vaccine only. In dose expansion phase, subjects will receive neoantigen tumor vaccine combination with PD-1/L1.
  Other Names: PGV002 mRNA Vaccine

SUMMARY:
This trial is an investigator-initiated, single-center, open-label, single-arm exploratory study of mRNA neoantigen tumor vaccine in the treatment of advanced gastric cancer, esophageal cancer, and liver cancer, including two phases: dose escalation and dose expansion. To evaluate the safety and tolerability of neoantigen tumor vaccine in subjects with advanced gastric cancer, esophageal cancer and liver cancer by conducting dose escalation trial in subjects diagnosed with advanced gastric cancer, esophageal cancer and liver cancer, and preliminarily evaluate the efficacy of neoantigen tumor vaccine in subjects with advanced gastric cancer, esophageal cancer and liver cancer. According to the characteristics of safety and efficacy data in the dose escalation phase, the dose expansion is performed at the intended clinical dose based on the investigator's judgment, and the treatment is performed in combination with PD-1/L1 to further evaluate the efficacy and safety profile of neoantigen tumor vaccine at a specific dose.

Both the dose escalation phase and dose expansion phase include a screening period (Week -4 ~ Week -2), a baseline period (Week -1 ~ Day -1), a treatment period (Day 1 ~ Week 8 or 16), and a follow-up period. Subjects who signed and provided the formal informed consent entered the screening period. The treatment period included the initial treatment period (Day 1 ~ Week 8) and the enhanced treatment period (Week 12 ~ Week 16). The investigator determined whether to enter the enhanced treatment period based on the comprehensive judgment of the subject's efficacy, safety, compliance and other factors from Week 8 to Week 12.

The dose escalation phase follows standard 3+3 design. 12-18 subjects are expected to be enrolled at 3 given dose level.

The investigator will choose the optimal clinical dose for dose expansion, which can be one dose group or multiple dose groups. PD-1/L1 drugs are used in parallel to further confirm the efficacy and safety of neoantigen tumor vaccine, with about 18 subjects. The usage and dosage of PD-1/L1 should aligned with the package insert.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and provided formal informed consent;
2. Male and female patients aged 18-75 years (inclusive);
3. Expected survival ≥ 3 months;
4. Subject with advanced gastric cancer, esophageal cancer and liver cancer proved by histopathology or cytology and who have failed to respond to standard treatment;
5. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors RECIST v1.1 (see Appendix 4, Response Evaluation Criteria in Solid Tumors) (i.e., mass ≥ 10 mm in diameter and malignant lymph node ≥ 15 mm in short diameter on enhanced spiral CT ≤ 5 mm);
6. ECOG performance status score of 0 ~ 2;
7. Treatment with other antineoplastic agents (e.g., chemotherapy, hormonal therapy, immunotherapy, antibody therapy, radiotherapy) for more than 5 half-lives of this agent or more than 4 weeks from baseline (whichever is shorter) during the baseline period ;
8. The organ function level must meet the following requirements (no blood transfusion or blood products, no hematopoietic stimulating factors, no albumin or blood products): absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count (PLT) ≥ 75 × 10^9/L, hemoglobin (Hb) ≥ 90 g/L; serum total bilirubin (TBIL) ≤ 1.5 ×ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN (if there is liver metastasis, total bilirubin ≤ 3 ×ULN, AST, ALT ≤ 5 ×ULN are allowed); Note: These laboratory tests may only be repeated once if the investigator deems it necessary (the reason for retest must be documented). If the criteria are met after retest, the laboratory parameter can be considered qualified.
9. Premenopausal women of childbearing potential must have a negative pregnancy test within 7 days prior to initiation of treatment and be non-lactating; women of non-childbearing potential are not required to have a pregnancy test and contraception unless participants are 50 years of age or older, have not used hormonal therapy and have been amenorrheic for at least 12 months, or have been surgically sterilized. All subjects (male or female) should use adequate barrier contraception throughout treatment and for 3 months after the end of treatment.

Exclusion Criteria:

1. Subject who need to receive systemic application of anti-allergic drugs for a long time, or have a history of life-threatening allergic reactions to any vaccine or drug;
2. Symptomatic or rapidly progressive central nervous system metastases. Patients with extensive lung metastases resulting in dyspnea; patients with tumors close to or invading major blood vessels or nerves;
3. New cerebrovascular accident (including ischemic stroke, hemorrhagic stroke, and transient ischemic attack) within 6 months before screening;
4. Subject with acute myocardial infarction within 6 months before screening, or uncontrolled angina, uncontrolled arrhythmia, severe heart failure (see Appendix 3, New York Heart Association Heart Failure Classification Criteria NYHA Class ≥ III) and other cardiovascular diseases;
5. Subject who have received treatment with immunomodulatory drugs 4 times before the first vaccination day (D1), including but not limited to: IL-2, CTLA-4 inhibitors, CD40 agonists, CD137 agonists, IFN-α (except for high-risk surgical subjects who use IFN-α as adjuvant therapy, if IFN-α treatment is stopped 4 times before this trial);
6. Subject with a history of renal insufficiency, serum creatinine level greater than 1.5 times the upper limit of normal;
7. Subject who received blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) before baseline;
8. Subject with skin diseases (e.g., psoriasis) at baseline that may prevent the intradermal injection of vaccine into the target area;
9. Subject still suffer from adverse reactions (except alopecia and platinum-induced neurotoxicity ≤ grade 2) that have not been restored to CTCAE version 5.0 grade ≤ 1 after previous anti-tumor treatment during the screening period;
10. Concomitant use of steroid hormone drugs (tumor or non-tumor related diseases) is required; however, topical application (not applied to the vaccination site) or inhaled steroid drugs are required;
11. Subject has an active infection or uncontrollable infection (except for simple urinary tract infection or upper respiratory tract infection) requiring systemic treatment; subjects with positive human immunodeficiency virus antibody, hepatitis B surface antigen and/or hepatitis B core antibody and positive hepatitis B virus deoxyribonucleic acid > 103 copies/mL, hepatitis C virus antibody, Treponema pallidum-specific antibody in virological monitoring during the screening period;
12. Hypertension poorly controlled on treatment (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
13. Subject with other malignant tumors within 5 years before the screening period, except for cervical carcinoma in situ, breast carcinoma in situ and cutaneous basal cell carcinoma that have received appropriate treatment and met the recovery criteria;
14. Subject with a history of autoimmune diseases [such as, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or hypothyroidism caused by chemoradiotherapy can be included), subjects with vitiligo or recovered asthma can be included without any intervention, and subjects with asthma requiring bronchodilators for medical intervention cannot be included];
15. Subject with active ulcer or gastrointestinal bleeding during the screening period;
16. Subject who has previously received similar therapeutic tumor vaccines;
17. Subject with congenital or acquired immunodeficiency;
18. Subject still participating in other clinical trials and not enrolled at the screening period;
19. Subject has a known alcohol or drug addiction;
20. Subject who is unable or unwilling to comply with the study protocol due to potential health, mental or social conditions in the opinion of the investigator;
21. Other conditions that, in the opinion of the investigator, would make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and degree of Adverse Events and Serious Adverse Events [Safety] | Up to 100 weeks
  Incidence and degree of participants with adverse events(CTCAE 5.0), abnormal laboratory tests (hematology, blood biochemistry, coagulation and urinalysis), abnormal ECG, abnormal echocardiography, abnormal vital signs and abnormal physical examination
Objective Response Rate (ORR) | Up to 100 weeks
  Objective Response Rate (ORR): The proportion of patients with complete response(CR) or partial response(PR) as measured by RECIST 1.1 criteria

SECONDARY OUTCOMES:
The establishment of recommended dose for further studies | Up to 16 weeks
  To determine the recommended dosage for pivotal study
Progression Free Survival (PFS) | Up to 100 weeks
  the time (in days) from the first dose of study treatment to the occurrence of disease progression; for subjects who die due to other causes before disease progression, the time (in days) from the date of entry into the treatment period to the date of death will be calculated, whichever occurs first. Response determination will be performed according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
The concentration of Serum cytokine | Up to 16 weeks
  IL-1β, IL-2, IL-6, IL-8, IL-10, TNF-α from time zero to time of last dose concentration
The concentration of Lymphocyte | Up to 16 weeks
  CD3+ 、CD3+∕CD4+ %、CD3+∕CD8+ %、CD4∕CD8 、CD3-∕CD19+ % from time zero to time of last dose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Dr., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No